CLINICAL TRIAL: NCT05678140
Title: The Effect of Instrument Assisted Soft Tissue Mobilization in Adhesive Capsulıtıs Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Basak Cigdem Karacay, Assistant professor, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-77504701-604.-02.
Record Dates: First submitted 2022-12-23; First posted 2023-01-10 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Adhesive Capsulitis; ınstrument assısted Soft tıssue molılızatıon
Keywords: adhesıve capsulıtis; ınstrument assısted soft tıssue molılızatıon
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: randomızed controlled trıal
Who Masked: Care Provider, Investigator
Masking Description: The researcher will not know which treatment is applied to the patients. The physiotherapist who gives the treatment will not know the results of the research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- soft tissue mobilization+conventional physical therapy (Experimental): Hot-pack to warm the superficial tissue, TENS for pain relief, ultrasound (US) to warm the joint structures before mobilization techniques, ROM, stretching, and isometric strengthening exercises to restore joint mobility and function of the shoulder area soft tissue mobilization; For the shoulder area, the application will take between 3-5 minutes. Instrumental Soft tissue mobilization will be performed while the participant is sitting in a supported chair, parallel to the shoulder and scapular muscle fibers and at an angle of 45 degrees to the vertical. Patients will be told that there may be small red spots called petechiae in the treated area. The application will be made using Graston iron rods.
  Interventions: Device: soft tissue mobilization; Other: conventional physical therapy
- conventional physical therapy (Placebo Comparator): Hot-pack to warm the superficial tissue, TENS for pain relief, ultrasound to warm the joint structures before mobilization techniques, ROM, stretching, and isometric strengthening exercises to restore joint mobility and function of the shoulder area.
  Interventions: Other: conventional physical therapy

INTERVENTIONS:
Device: soft tissue mobilization — soft tissue mobilization; For the shoulder area, the application will take between 3-5 minutes. Instrumental Soft tissue mobilization will be performed while the participant is sitting in a supported chair, parallel to the shoulder and scapular muscle fibers and at an angle of 45 degrees to the vertical. Patients will be told that there may be small red spots called petechiae in the treated area. The application will be made using Graston iron rods.
  Arms: soft tissue mobilization+conventional physical therapy
Other: conventional physical therapy — Hot-pack to warm the superficial tissue, TENS for pain relief, ultrasound (US) to warm the joint structures before mobilization techniques, ROM, stretching, and isometric strengthening exercises to restore joint mobility and function of the shoulder area

SUMMARY:
The primer aim of this study is to demonstrate the effect of instrument assisted soft tissue mobılızatıon on paın ,functıonality, joint range of motion patients with adhesive capsulitis

DETAILED DESCRIPTION:
Adhesive capsulitis is also called arthrofibrosis, which involves excessive adhesion formation along the glenohumeral joint. It is a disease of unknown etiology and is classified as primary and secondary. Primary adhesive capsulitis includes cases of idiopathic origin resulting from chronic inflammation with fibroblast proliferation. Secondary adhesive capsulitis, central nervous system involvement, arm immobilized for a long time, trauma or fracture, infectious diseases, etc. Includes post-mortem situations.

It is characterized by shoulder pain, decreased range of motion, and limitation of function. This affects the function of the entire upper extremity. Idiopathic adhesive capsulitis usually involves the non-dominant upper extremity, with bilateral involvement in 40-50% of cases. It is more common in women between the ages of 40 and 60. The incidence of adhesive capsulitis among the population is between 3% and 5%. It has been reported with up to 20% higher incidence in the diabetic population. It is also associated with other pathological disorders such as thyroid dysfunction, coronary artery disease and cerebrovascular disease. Although the pathology is self-limiting, long-term symptoms develop in approximately 20% to 50% of cases.

Adhesive capsulitis progression is characterized by four stages, each stage presenting a distinctive clinical picture.

1. The painful phase lasts less than three months and presents with shoulder pain at night when glenohumeral movement is preserved.
2. The freezing process lasts three to nine months and is manifested by severe pain and stiffness in the glenohumeral joint.
3. The frozen shoulder process lasts nine to fourteen months and is eventually characterized by loss of motion and pain in all directions.
4. The resolution phase lasts for fifteen to twenty-four months and is characterized by persistent stiffness, minimal pain, and delayed improvement in shoulder motion.

Abnormal shoulder kinematics develops in response to the lack of extensibility of the capsule with the change in motor patterns in the central nervous system. Increased thoracic kyphosis can be seen as postural deviations. However, fibrotic changes are also seen in the periarticular connective tissue and trigger points. This presents as a higher level of disability with painful shoulder. Physiotherapy is the mainstay of treatment for patients with adhesive capsulitis. Joint mobilization has a proven role in conjunction with Codman's exercises. Transcutaneous Electrical Nerve Stimulation (TENS), Diathermy is used in the treatment to reduce pain. Instrument Assisted Soft Tissue Mobilization (IASTM) is a soft tissue mobilization method that works by generating localized inflammation and facilitates collagen synthesis and realignment. In fact, when IASTM is given to soft tissues with appropriate pressure, localized inflammation occurs with microvascular bleeding. This will increase blood flow to the injured area along with the recruitment of more fibroblasts. With the removal of scar tissues and adhesions, healing will be supported by the organization of collagen of fibroblasts. The fibronectin induced by IASTM is required for tissue repair. A localized force will be transmitted through an instrument to the affected tissues to leave a scar.

IASTM has become increasingly popular as a tool for the rehabilitation of sports injuries. It has been proven to be successful in a short time in reducing pain and increasing mobility after sports injuries. There are studies showing an increase in ROM after a single application of this technique.

It is known that it takes a long time to relieve pain and achieve a good improvement in ROM in adhesive capsulitis. This affects their quality of life and creates the need for treatment options that provide a shorter recovery time. Various conservative protocols are followed with physical therapy as the main treatment in adhesive capsulitis. Few studies have used IASTM as a treatment to evaluate its effect on adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

- 1.Male and Female patients aged 20-60 years 2.Diagnosed with adhesive capsulitis 2. Loss of range of motion in the capsular pattern (external rotation > abduction > internal rotation) will be included in the study.

3. consent to participate

Exclusion Criteria:

* 1. Injury to the upper extremity in the last 6 months 2. Shoulder injection in the last 6 months 3. Existing open wound in the upper extremity area 4. Previous upper extremity surgery 5. Being hypersensitive 6. Having a generalized infection 7. Having uncontrolled hypertension 8. Inability to cooperate; 9. The patient's unwillingness to participate in the study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | baseline
  Visual Analogue Scale (VAS) for pain assesment .In tgis scale ,evaluaments paın with 10- point Likert scale , 0 is scored as no pain,5 as modarete pain , and 10 as excrucıatıng pain.
Visual Analogue Scale (VAS) | 2. week (in the middle of treatment)
  Visual Analogue Scale (VAS) for pain assesment .In tgis scale ,evaluaments paın with 10- point Likert scale , 0 is scored as no pain,5 as modarete pain , and 10 as excrucıatıng pain.
Visual Analogue Scale (VAS) | 4. week (at the end of treatment)
  Visual Analogue Scale (VAS) for pain assesment .In tgis scale ,evaluaments paın with 10- point Likert scale , 0 is scored as no pain,5 as modarete pain , and 10 as excrucıatıng pain.
The Shoulder Pain and Disability Index (SPADI) | baseline
  SPADI is a pain and functional disability questionnaire specifically for the shoulder. It is divided into two parts: the pain scale (5 questions) and the disability scale (8 questions). Each question is rated on a scale from 0 to 10. The final score is calculated as a percentage.
The Shoulder Pain and Disability Index (SPADI) | 2. week (in the middle of treatment)
  SPADI is a pain and functional disability questionnaire specifically for the shoulder. It is divided into two parts: the pain scale (5 questions) and the disability scale (8 questions). Each question is rated on a scale from 0 to 10. The final score is calculated as a percentage.
The Shoulder Pain and Disability Index (SPADI) | 4. week (at the end of treatment)
  SPADI is a pain and functional disability questionnaire specifically for the shoulder. It is divided into two parts: the pain scale (5 questions) and the disability scale (8 questions). Each question is rated on a scale from 0 to 10. The final score is calculated as a percentage.

SECONDARY OUTCOMES:
joint range of motion | baseline
  measured using a protractor. Shoulder flexion, extension, abduction, internal rotation and external rotation intervals are measured in the supine position.
joint range of motion | 2. week (in the middle of treatment)
  measured using a protractor. Shoulder flexion, extension, abduction, internal rotation and external rotation intervals are measured in the supine position.
joint range of motion | 4. week (at the end of treatment)
  measured using a protractor. Shoulder flexion, extension, abduction, internal rotation and external rotation intervals are measured in the supine position.

CONTACTS AND LOCATIONS:
Overall Officials: Basak Cigdem Karacay, Assoc. Prof, Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kırşehir Ahi Evran University Faculty of Medicine, Kırşehir, City Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aggarwal A, Saxena K, Palekar TJ, Rathi M. Instrument assisted soft tissue mobilization in adhesive capsulitis: A randomized clinical trial. J Bodyw Mov Ther. 2021 Apr;26:435-442. doi: 10.1016/j.jbmt.2020.12.039. Epub 2020 Dec 31. PMID 33992280
- [Result] Laudner K, Compton BD, McLoda TA, Walters CM. Acute effects of instrument assisted soft tissue mobilization for improving posterior shoulder range of motion in collegiate baseball players. Int J Sports Phys Ther. 2014 Feb;9(1):1-7. PMID 24567849
- [Result] Hussey MJ, Boron-Magulick AE, Valovich McLeod TC, Welch Bacon CE. The Comparison of Instrument-Assisted Soft Tissue Mobilization and Self-Stretch Measures to Increase Shoulder Range of Motion in Overhead Athletes: A Critically Appraised Topic. J Sport Rehabil. 2018 Jul 1;27(4):385-389. doi: 10.1123/jsr.2016-0213. Epub 2018 Jun 1. PMID 28253058